CLINICAL TRIAL: NCT07407283
Title: A Multicenter, Open-label, Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of SHR-4394 in Combination With Anti-tumor Therapy in Participants With Prostate Cancer
Brief Title: A Clinical Study of SHR-4394 in Combination With Anti-tumor Therapy in Prostate Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4394-201
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tazemetostat

STUDY DESIGN:
Intervention Model Description: SHR-4394 in combination with anti-tumor therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-4394 in combination with anti-tumor therapy Group (Experimental): SHR-4394, Rezvilutamide, HRS-5041, Tazemetostat.
  Interventions: Drug: SHR-4394; Drug: Rezvilutamide; Drug: HRS-5041 Tablets; Drug: Tazemetostat

INTERVENTIONS:
Drug: SHR-4394 — SHR-4394.
Drug: Rezvilutamide — Rezvilutamide tablets.
Drug: HRS-5041 Tablets — HRS-5041 tablets.
Drug: Tazemetostat — Tazemetostat tablets.

SUMMARY:
The study aims to assess the safety and tolerability of SHR-4394 in combination with anti-tumor therapy in participants with prostate cancer, and determine the recommended Phase II dose (RP2D); To evaluate of the efficacy of SHR-4394 in combination with anti-tumor therapy in participants with prostate cancer based on Prostate-Specific Antigen (PSA) response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 85 years (inclusive) at the time of signing the informed consent form (with an upper age limit of 80 years for the dose escalation phase), and male.
2. Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Life expectancy is expected to be at least 12 weeks.
4. Must have a prostate-specific antigen (PSA) level of ≥1 ng/mL during the screening period.
5. Ongoing therapy with a luteinizing hormone-releasing hormone analog (LHRHa) for medical castration or prior bilateral orchiectomy for surgical castration; participants who have not undergone bilateral orchiectomy must plan to maintain effective LHRHa therapy throughout the study period.
6. Must have histologically or cytologically confirmed prostate adenocarcinoma, without a diagnosis of neuroendocrine carcinoma or small cell carcinoma.
7. Must have radiographically confirmed metastatic disease by CT/MRI or radionuclide bone scan (⁹⁹ᵐTc).
8. Male participants with female partners of childbearing potential must practice highly effective contraception from the time of signing the informed consent form until 5 months after the last dose of the investigational product, and must refrain from donating sperm during this period.

Exclusion Criteria:

1. Planning to receive any other anti-tumor therapy during the course of this study.
2. Have received any other investigational drugs or treatments not yet approved for marketing within 4 weeks prior to the first dose in this study.
3. Have undergone surgery requiring endotracheal intubation and general anesthesia within 28 days prior to the first dose, minor diagnostic or superficial surgery within 7 days prior to the first dose, or are scheduled to undergo elective surgery during the trial period.
4. Have not recovered from adverse events due to prior anti-tumor therapy to ≤ Grade 1 according to NCI-CTCAE v6.0 (with the exception of Grade 2 peripheral neuropathy, alopecia, hypothyroidism controlled with hormone replacement therapy, and well-controlled type 1 diabetes managed with insulin).
5. Known history of hypersensitivity to the investigational drug(s) to be used or any of their excipients.
6. Participants with untreated or inadequately treated central nervous system (CNS) metastases, or uncontrolled or symptomatic active CNS metastases are excluded. However, participants may be eligible if their CNS metastases have been adequately treated, and any neurological symptoms have resolved or been stable for at least 4 weeks prior to enrollment (residual signs or symptoms related to the CNS treatment are allowed).
7. Uncontrolled tumor-related pain, as determined by the investigator. Participants requiring analgesic medication must be on a stable analgesic regimen at the time of study entry.
8. Presence of uncontrolled third-space effusions (e.g., pleural effusion, pericardial effusion, or ascites) that, despite therapeutic interventions such as drainage within 28 days prior to the first dose, remain uncontrolled or rapidly recur after drainage, requiring repeated drainage procedures.
9. History of any other malignancy within 5 years prior to the first dose, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin, radically resected papillary thyroid carcinoma, and radically resected ductal carcinoma in situ of the breast.
10. History of epilepsy or any condition predisposing to seizures (such as transient ischemic attack, stroke, or traumatic brain injury with loss of consciousness requiring hospitalization) within 12 months prior to enrollment.
11. History of interstitial pneumonia (ILD) or interstitial lung disease (including cases requiring steroid therapy), or any other history of pulmonary fibrosis, organizing pneumonia, drug- or radiation-induced pneumonitis, congenital pneumonitis, or any evidence of active pneumonia on chest CT scan that may interfere with the assessment of immune-related pulmonary toxicity.
12. Active severe gastrointestinal disorders, including but not limited to complete or incomplete bowel obstruction, persistent/recurrent diarrhea (or diarrhea with fever), moderate to severe gastrointestinal hemorrhage (including endoscopically active bleeding), gastric or duodenal ulcers, gastrointestinal perforation, acute pancreatitis, ulcerative colitis, congenital megacolon, Crohn's disease, etc.
13. Exclusion is required for: a history of severe infection within 4 weeks prior to the first dose; active infection requiring systemic antibiotics within 2 weeks prior to the first dose; or evidence of active tuberculosis infection within 1 year prior to enrollment. A history of active tuberculosis (TB) infection more than 1 year ago without adequate treatment is also excluded.
14. Active hepatitis B virus or hepatitis C virus (HBV/HCV) infection (HBsAg+ with DNA ≥ 2000 IU/mL; HCV Ab+ with RNA > ULN).
15. Participants are excluded if they have a history of immunodeficiency (including HIV positivity, other acquired or congenital immunodeficiencies) or organ transplantation, or a history of active autoimmune disease. Exceptions include participants with immune disorders not requiring systemic treatment (e.g., vitiligo, psoriasis) or autoimmune conditions well-controlled by hormone replacement therapy (e.g., type 1 diabetes, hypothyroidism).
16. History of severe cardiovascular or cerebrovascular disease.
17. History of arterial or venous thromboembolic events within 3 months prior to the first dose, or the presence of arterial/venous thrombosis (e.g., deep vein thrombosis, pulmonary embolism) identified during screening.
18. Any concomitant illness, condition, or social circumstance that, in the judgment of the investigator, could compromise participant safety or interfere with the completion of the study.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of SHR-4394 combined with anti-tumor therapy in prostate cancer participants | About 12 months.
  Phase I.
The incidence and severity of adverse events (AEs) | About 12 months.
  Phase I.
Prostate-Specific Antigen response rate (PSA50) | About 16 months.
  Phase II.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | About 28 months.
  Efficacy endpoints of SHR-4394 in combination with anti-tumor therapy in participants with prostate cancer.
Disease Control Rate (DCR) | About 28 months.
  Efficacy endpoints of SHR-4394 in combination with anti-tumor therapy in participants with prostate cancer.
Duration of Response (DoR) | About 28 months.
  Efficacy endpoints of SHR-4394 in combination with anti-tumor therapy in participants with prostate cancer.
Prostate-Specific Antigen (PSA) Response Rate | About 28 months.
  Efficacy endpoints of SHR-4394 in combination with anti-tumor therapy in participants with prostate cancer.
Time to PSA progression | About 28 months.
  Efficacy endpoints of SHR-4394 in combination with anti-tumor therapy in participants with prostate cancer.
Radiographic Progression-Free Survival (rPFS) | About 28 months.
  Efficacy endpoints of SHR-4394 in combination with anti-tumor therapy in participants with prostate cancer.
Overall Survival (OS) | About 28 months.
  Efficacy endpoints of SHR-4394 in combination with anti-tumor therapy in participants with prostate cancer.
Plasma concentrations of SHR-4394 and its combination drugs | About 12 months.
  Phase I.
Prostate-Specific Antigen response rate (PSA90) | About 28 months.
  Phase II.
Proportion of participants with undetectable PSA | About 6 months.
  Phase II.
Incidence and severity of adverse events (AEs) | About 16 months.
  Phase II.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided